CLINICAL TRIAL: NCT05840952
Title: A First-in-Human Multi-Part Phase 1 Study in Healthy Volunteers to Evaluate the Safety, Tolerability, Pharmacokinetics, and Drug-Drug Interaction Potential of Single and Multiple Doses of ALG-097558
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aligos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALG-097558-701
Record Dates: First submitted 2023-04-10; First posted 2023-05-03 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-09

CONDITIONS: COVID-19
Keywords: Healthy Volunteer
MeSH Terms: conditions — COVID-19 | interventions — Midazolam; Itraconazole; Carbamazepine

STUDY DESIGN:
Intervention Model Description: Parts 1 and 2 of the study are parallel assignment, with 2 arms. Parts 3, 5, and 6 are fixed sequence, crossover studies. Part 4 is a partially placebo-controlled, fixed sequence, crossover study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Parts 1 and 2 are double blinded and randomized. Parts 3, 5, and 6 are open label and non-randomized. Part 4 is partially singled blinded non-randomized. Participants are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- ALG-097558 (Experimental): Oral doses of ALG-097558 in Healthy Volunteers, up to 20 doses over 10 days
  Interventions: Drug: ALG-097558
- Placebo (Placebo Comparator): Oral doses of placebo in Healthy Volunteers, up to 20 doses over 10 days
  Interventions: Drug: Placebo
- ALG-097558 and Midazolam (Experimental): Oral doses of ALG-097558, up to 14 doses over 7 days and oral dose of Midazolam, up to 2 doses, over 2 days, in Healthy Volunteers
  Interventions: Drug: ALG-097558; Drug: Midazolam
- ALG-097558, Placebo, and, Itraconazole (Experimental): Oral doses of placebo, up to 2 doses over 2 days, followed by ALG-097558, up to 2 doses over 2 days, and itraconazole up to 10 doses over 10 days, in Healthy Volunteers.
  Interventions: Drug: ALG-097558; Drug: Placebo; Drug: Itraconazole
- ALG-097558 and Carbamazepine (Experimental): Oral doses of ALG-097558, up to 2 doses over 2 days and oral doses of Carbamazepine, up to 30 doses, over 15 days, in Healthy Volunteers
  Interventions: Drug: ALG-097558; Drug: Carbamazepine
- ALG-097558 Bioavailability (Experimental): Oral doses of ALG-097558, up to 3 doses over 3 days, both solution and tablet formulations dosed in fasted state, and tablet formulation dosed in fed state, in Healthy Volunteers
  Interventions: Drug: ALG-097558 in solution formulation; Drug: ALG-097558 in tablet formulation

INTERVENTIONS:
Drug: ALG-097558 — single or multiple doses of ALG-097558
  Arms: ALG-097558; ALG-097558 and Carbamazepine; ALG-097558 and Midazolam; ALG-097558, Placebo, and, Itraconazole
Drug: Placebo — single or multiple doses of placebo
  Arms: ALG-097558, Placebo, and, Itraconazole; Placebo
Drug: Midazolam — Multiple doses of Midazolam
  Arms: ALG-097558 and Midazolam
Drug: Itraconazole — Multiple doses of Itraconazole
  Arms: ALG-097558, Placebo, and, Itraconazole
Drug: Carbamazepine — Multiple doses of Carbamazepine
  Arms: ALG-097558 and Carbamazepine
Drug: ALG-097558 in solution formulation — ALG-097558 in solution administered in fasted state
  Arms: ALG-097558 Bioavailability
Drug: ALG-097558 in tablet formulation — ALG-097558 in tablet administered in fasted and fed state
  Arms: ALG-097558 Bioavailability

SUMMARY:
A multi-part study of ALG-097558 to evaluate safety, tolerability, pharmacokinetics and drug-drug interaction potential after single and multiple doses in healthy volunteers

ELIGIBILITY:
Inclusion Criteria for All Subjects:

1. Male and Female between 18 and 55 years old
2. BMI 18.0 to 32.0 kg/m^2
3. Female subjects must have a negative serum pregnancy test at screening
4. Subjects must have a 12-lead electrocardiogram (ECG) that meets the protocol criteria

Exclusion Criteria for All Subjects:

1. Subjects with any current or previous illness that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject or that could prevent, limit, or confound the protocol specified assessments or study results' interpretation
2. Subjects with a past history of cardiac arrhythmias, risk factors for Torsade de Pointes syndrome (e.g., hypokalemia, family history of long QT Syndrome) or history or clinical evidence at screening of significant or unstable cardiac disease etc.
3. Subjects with a history of clinically significant drug allergy
4. Excessive use of alcohol defined as regular consumption of ≥14 units/week
5. Unwilling to abstain from alcohol use for 1 week prior to start of the study through end of study follow up
6. Subjects with Hepatitis A, B, C, E or HIV-1/HIV-2 infection or acute infections such as SARS- CoV-2 infection
7. Subjects with renal dysfunction (e.g., estimated creatinine clearance <90 mL/min/1.73 m^2 at screening, calculated by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 11 days for Part 1
  The number and severity of treatment emergent adverse events as assessed by DAIDS v2.1
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 20 days for Part 2
  The number and severity of treatment emergent adverse events as assessed by DAIDS v2.1
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 20 days for Part 3
  The number and severity of treatment emergent adverse events as assessed by DAIDS v2.1
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 23 days for Part 4
  The number and severity of treatment emergent adverse events as assessed by DAIDS v2.1
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 28 days for Part 5
  The number and severity of treatment emergent adverse events as assessed by DAIDS v2.1
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 17 days for Part 6
  The number and severity of treatment emergent adverse events as assessed by DAIDS v2.1
Area under the concentration time curve [AUC] | Predose (-2 hours) up to 11 days
  Pharmacokinetic parameters of Midazolam and applicable metabolites
Time to maximum plasma concentration [Tmax] | Predose (-2 hours) up to 11 days
  Pharmacokinetic parameters of Midazolam and applicable metabolites
Maximum plasma concentration [Cmax] | Predose (-2 hours) up to 11 days
  Pharmacokinetic parameters of Midazolam and applicable metabolites
Minimum plasma concentration [Cmin] | Predose (-2 hours) up to 11 days
  Pharmacokinetic parameters of Midazolam and applicable metabolites
C0 [predose] | Predose (-2 hours) up to 11 days
  Pharmacokinetic parameters of Midazolam and applicable metabolites
Half-life [t1/2] | Predose (-2 hours) up to 11 days
  Pharmacokinetic parameters of Midazolam and applicable metabolites
Area under the concentration time curve [AUC] | Predose (-0.75 hours) up to 19 days
  Pharmacokinetic parameters of ALG-07558 and metabolite ALG-097730 following administration of itraconazole or carbamazepine
Time to maximum plasma concentration [Tmax] | Predose (-0.75 hours) up to 19 days
  Pharmacokinetic parameters of ALG-07558 and metabolite ALG-097730 following administration of itraconazole or carbamazepine
Maximum plasma concentration [Cmax] | Predose (-0.75 hours) up to 19 days
  Pharmacokinetic parameters of ALG-07558 and metabolite ALG-097730 following administration of itraconazole or carbamazepine
Minimum plasma concentration [Cmin] | Predose (-0.75 hours) up to 19 days
  Pharmacokinetic parameters of ALG-07558 and metabolite ALG-097730 following administration of itraconazole or carbamazepine
C0 [predose] | Predose (-0.75 hours) up to 19 days
  Pharmacokinetic parameters of ALG-07558 and metabolite ALG-097730 following administration of itraconazole or carbamazepine
Half-life [t1/2] | Predose (-0.75 hours) up to 19 days
  Pharmacokinetic parameters of ALG-07558 and metabolite ALG-097730 following administration of itraconazole or carbamazepine
Area under the concentration time curve [AUC] | Predose (-0.75 hours) up to 9 days
  Pharmacokinetic parameters of ALG-07558 and metabolite ALG-097730 following administration of ALG-097558 in either solution or tablet formulations and following a high fat diet
Time to maximum plasma concentration [Tmax] | Predose (-0.75 hours) up to 9 days
  Pharmacokinetic parameters of ALG-07558 and metabolite ALG-097730 following administration of ALG-097558 in either solution or tablet formulations and following a high fat diet
Maximum plasma concentration [Cmax] | Predose (-0.75 hours) up to 9 days
  Pharmacokinetic parameters of ALG-07558 and metabolite ALG-097730 following administration of ALG-097558 in either solution or tablet formulations and following a high fat diet
Minimum plasma concentration [Cmin] | Predose (-0.75 hours) up to 9 days
  Pharmacokinetic parameters of ALG-07558 and metabolite ALG-097730 following administration of ALG-097558 in either solution or tablet formulations and following a high fat diet
C0 [predose] | Predose (-0.75 hours) up to 9 days
  Pharmacokinetic parameters of ALG-07558 and metabolite ALG-097730 following administration of ALG-097558 in either solution or tablet formulations and following a high fat diet
Half-life [t1/2] | Predose (-0.75 hours) up to 9 days
  Pharmacokinetic parameters of ALG-07558 and metabolite ALG-097730 following administration of ALG-097558 in either solution or tablet formulations and following a high fat diet

SECONDARY OUTCOMES:
Maximum plasma concentration [Cmax] | Predose (-0.75 hours) up to 19 days
  Pharmacokinetic parameters of ALG-097558 in plasma
Area under the concentration time curve [AUC] | Predose (-0.75 hours) up to 19 days
  Pharmacokinetic parameters of ALG-097558 in plasma
Time to maximum plasma concentration [Tmax] | Predose (-0.75 hours) up to 19 days
  Pharmacokinetic parameters of ALG-097558 in plasma
Minimum plasma concentration [Cmin] | Predose (-0.75 hours) up to 19 days
  Pharmacokinetic parameters of ALG-097558 in plasma
Half-life [t1/2] | Predose (-0.75 hours) up to 19 days
  Pharmacokinetic parameters of ALG-097558 in plasma
C0 [predose] | Predose (-0.75 hours) up to 19 days
  Pharmacokinetic parameters of ALG-097558 in plasma
Dose Proportionality | Predose (-0.75 hours) up to 19 days
  Pharmacokinetic parameters of ALG-097558 in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No